CLINICAL TRIAL: NCT02202070
Title: Phase 1 Study of Role of Botox in Myofascial Temporomandibular Disorder
Brief Title: Botox for Treatment of TMJ Disorder With Bruxism
Acronym: TMJ
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ethan Baughman, Plastic surgery resident physician, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AAHEJB
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Temporomandibular Joint Disorders; Bruxism; Temporomandibular Joint Dysfunction Syndrome; Myofascial Pain Dysfunction Syndrome, Temporomandibular Joint
Keywords: onabotulinumtoxinA; Temporomandibular Joint Disorders; Bruxism; Temporomandibular Joint Dysfunction Syndrome; Myofascial Pain Dysfunction Syndrome, Temporomandibular Joint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism; Temporomandibular Joint Dysfunction Syndrome | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox injection first, followed by placebo (Experimental): 50 units Botox injection in masseter and temporalis muscles in the first 3 months, then second injection of normal saline at placebo in second 3 months
  Interventions: Drug: onabotulinumtoxinA
- Placebo injection first, followed Botox (Experimental): Injection of normal saline at placebo in first 3 months, then 50 units Botox injection in masseter and temporalis muscles in the second 3 months.
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA
  Other Names: BOTOX

SUMMARY:
Hypothesis: Myofascial temporomandibular joint disorder and related symptoms are associated with mandibular condyle and temporal fossa overloading secondary to temporalis and masseter muscle hyperactivity and spasm

This study will examine the use of onabotulinumtoxinA (Botox) to treat myofascial pain disorder in patients with bruxism who frequently exhibit signs of temporomandibular joint disorder (TMD) in a double blind cross-over randomized clinical trial by injecting 50 units Botox in temporalis and masseter muscles in 32 patients with 6 months follow up.

The objective of the proposed study will be to establish the safety and efficacy of botox in treating TMD associated with bruxism. By the time patients reach the specialists office, most have failed maximal conservative therapies, including non-chew diet, night guard, oral analgesics, muscle relaxants, physical therapy, and a portion have even undergone more invasive procedures, such as manipulation under anesthesia, arthroscopy, and arthroplasty surgeries with limited improvement or recurrence. Primary outcome of the study will be 50% reduction in pain. Secondary outcomes will be 50% reduction in surgical therapy, 25% increase in maximal inter-incisal opening (MIO). The investigators look forward to working with you on the proposed study

DETAILED DESCRIPTION:
The study will enroll 32 patients with myofascial TMD. Patient will be aged 18-65. Exclusion criteria will include neuromuscular diseases, prior botox injections within previous 12 months, pregnancy, and fibromyalgia. All patients will be selected from the outpatient clinic, complaining of TMJ disease associated with bruxism. Screening will include a thorough history and exam, and TMJ CT scan or MRI. Patients with neuromuscular disorders, musculoskeletal disorders, and prior Botox injections will be excluded. Patients who have not already undergone conservative treatment will be managed with 3 months conservative therapies prior to becoming eligible. All patients will be informed and consented for participation in the study and Botox injections. Baseline pain questionnaire, physical exam will be performed. Patients will be randomized to receive normal saline or botox injections. All patients will crossover for the second set of injections at 3 months. All patients will receive up to a total of 200 Botox units at either 0 or 3 month time points. In this regard, patients will act as their own placebo control. Botox will be prepared according to the manufacturer's instructions. Briefly, the lyophilized protein will be reconstituted with preservative-free normal saline and drawn into 1-mL syringe. While the patient is sitting in the office procedure chair, 25 to 50 U of Botox will be injected into each temporalis muscle and 25 to 50 U of Botox will be injected into the each masseter muscle. The patient will be instructed to keep head elevated for 8 hours. Patients will be called 3 times after the first round of injections, to monitor for adverse events. Patients will be seen in clinic at 3 months and asked to fill out a second pain questionnaire. They will also undergo second physical exam, and then receive a second set of injections (crossover). Patients will be seen in clinic at 6 months and asked to fill out a third pain questionnaire undergo third physical exam. Patients will be called 3 times after the second round of injections, to monitor for adverse events. Patients will be seen in clinic at 6 months and asked to fill out a third pain questionnaire undergo a third physical exam

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 persons with a diagnosis of myofascial temporomandibular joint disorder refractory to conservative treatment for 6 months

Exclusion Criteria:

* pregnancy
* rheumatoid arthritis
* ankylosing spondylitis
* psoriatic arthritis
* fibromyalgia
* neuropathic pain
* pain of dental origin
* muscle relaxant use
* aminoglycoside use
* prior Botox use
* neuropathic pain
* trigeminal neuralgia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
50% reduction in pain | 6 months
  Patients will be seen in clinic every 3 months and asked to fill out questionaire. Questionaire will include with visual analogue scale (VAS) average pain over previous week, month

SECONDARY OUTCOMES:
25% increase in maximal opening at incisors | 6 months
  Patients will be seen in clinic every 3 months. Providers will objectively measure maximal opening at incisors (MOI), lateral and anterior mandible excursion on clinical exam.

OTHER OUTCOMES:
50% reduction in progression of disease to surgery | 6 months
  Patients will be monitored for TMJ arthoscopic and arthoplasty procedures

CONTACTS AND LOCATIONS:
Overall Officials: Alan A Harvey, DMD, Principal Investigator — Assistant Professor, Department of Otolaryngology
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States